CLINICAL TRIAL: NCT01578057
Title: A Randomized, Double-mask, Four-period Crossover Study in Healthy Subjects to Evaluate the Pharmacodynamic and Pharmacokinetic Interactions of Tasimelteon and Ethanol
Brief Title: Evaluation of the Pharmacodynamic and Pharmacokinetic Interactions of Tasimelteon and Ethanol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1108
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Pharmacodyamics and Pharmacokinetics of Tasimelteon Alone and in Combination With Ethanol
Keywords: alcohol
MeSH Terms: interventions — tasimelteon; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- tasimelteon + placebo ethanol (Experimental)
  Interventions: Drug: tasimelteon; Drug: Placebo ethanol
- ethanol + placebo tasimelteon (Experimental)
  Interventions: Drug: Ethanol; Other: Placebo tasimelteon
- tasimelteon + ethanol (Experimental)
  Interventions: Drug: tasimelteon; Drug: Ethanol
- placebo tasimelteon + placebo ethanol (Experimental)
  Interventions: Other: Placebo tasimelteon; Drug: Placebo ethanol

INTERVENTIONS:
Drug: tasimelteon — 20mg, once
  Other Names: VEC-162; BMS-214778
  Arms: tasimelteon + ethanol; tasimelteon + placebo ethanol
Drug: Ethanol — 0.6 g/kg ethanol (women) or 0.7 g/kg ethanol (men) in a total volume of 300 mL as a light cranberry juice cocktail, (consumed within 15 minutes).
  Other Names: vodka
  Arms: ethanol + placebo tasimelteon; tasimelteon + ethanol
Other: Placebo tasimelteon — once
  Arms: ethanol + placebo tasimelteon; placebo tasimelteon + placebo ethanol
Drug: Placebo ethanol — A total volume of 300 mL as a light cranberry cocktail (consumed within 15 minutes) with about 1 mL of supernatant of ethanol in the top
  Arms: placebo tasimelteon + placebo ethanol; tasimelteon + placebo ethanol

SUMMARY:
The purpose of this research study is to understand if there is any difference in the effects of tasimelteon when it is taken alone or in combination with alcohol. This research study is also being done to understand if there is any difference in the amount of tasimelteon (and its breakdown products) or alcohol in the blood when taken alone or together. Finally, the study will also look at the safety and tolerability (how acceptable it is) of tasimelteon.

DETAILED DESCRIPTION:
Alcohol is a drug that gets absorbed into the bloodstream quickly. The blood carries the alcohol to the brain where it slows down the messages in the brain (alcohol is a depressant). Alcohol affects a person's memory, behaviour, concentration, alertness (your thought process is slower), and coordination (your movements become clumsy). The intended effect of tasimelteon is to cause sleepiness. Sleepiness may result in similar effects on memory, concentration, alertness, and coordination as alcohol. There is the possibility taking tasimelteon and alcohol together can make these effects stronger or worse.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and acceptance to provide written informed consent;
2. Men or women between 19- 75 years, inclusive;
3. Subjects with Body Mass Index (BMI) of ≥18.0 and ≤35.0 kg/m2 (BMI = weight (kg)/ [height (m)]2) and weigh a minimum of 50 kg (110 pounds);
4. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing and females must have a negative pregnancy test at the screening and baseline visits; Note: Acceptable methods of birth control include any one of the following: abstinence, vasectomized sexual partner, hormonal methods (i.e. pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam.
5. Social or moderate drinkers who drink on average 7 to 21 units of alcohol per week and have consumed more than 4 (women) or 5 (men) units of alcohol on at least one occasion in the last month; Note: One unit of alcohol is equivalent to 1.5 oz of hard liquor or 5 oz of wine or 12 oz of beer.
6. Willing and able to comply with study requirements and restrictions;
7. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;
8. Vital signs (after 3 minutes resting in a semi-supine or seated position) which are within the ranges shown below:

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 90-150 mm Hg;
   3. Diastolic blood pressure between 50-95 mm Hg;
   4. Pulse rate between 40-100 bpm.

Exclusion Criteria:

1. Subjects who are not able to tolerate [0.6 g/kg for female/0.7 g/kg for men] ethanol during the Qualification visit. Intolerance is defined as ≥ 1 vomiting episode or severe nausea.
2. Current (within 12 months) drug or alcohol abuse or dependence as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse or evidence of such abuse as indicated by the laboratory assays conducted during the Screening Visit or at Baseline;
3. Any major surgery within three months of Baseline or any minor surgery within one month;
4. History or current evidence of pulmonary, cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction judged by the Investigator to be clinically significant;
5. Subjects who are currently considered a suicide risk, any subject who has ever made a suicide attempt, or those who are currently demonstrating active (within the last year) suicidal ideation as deemed by the Columbia Suicide Severity Rating Scale (C-SSRS);
6. Any condition requiring the regular use of medication;
7. Subjects who have used tobacco products 3 months prior to Baseline. Smokers will be defined as any subject who reports cigarette, tobacco, nicotine gum, or nicotine patch use;
8. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of Baseline;
9. Donation or loss of 400 mL or more of blood within two months prior to the Baseline Visit;
10. Significant illness within the two weeks prior to Baseline;
11. A known intolerance or hypersensitivity to tasimelteon or drugs similar to tasimelteon including melatonin;
12. Pregnant or lactating females;
13. History of liver disease and/or positive for one or more of the following serological results:

    1. A positive hepatitis B surface antigen (HBsAg)
    2. A positive hepatitis C antibody test (anti-HCV)
    3. A positive HIV test result;
14. Use of prescription or OTC medication, including melatonin and herbal products (e.g., St. John's Wort) within 2 weeks of the Baseline Visit;
15. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 day preceding the Screening visit;
16. Participation in a previous BMS-214778/VEC-162 trial;
17. Inability to be venipunctured and/or tolerate venous access;
18. Subjects who are unable to read or speak English;
19. Any other sound medical reason as determined by the clinical Investigator.

Ages: 19 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameters (Digit Vigilance, Digit Symbol Substitution Task, Hopkins Verbal Learning Test Revised , Divided Attention Test, Balance Platform Test, Choice Reaction Time, Visual Analog Scale) as measured by peak change from baseline | Days 1, 8, 15, 22: at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours after dose
  Differences will be calculated for the following comparisons:
  * Ethanol Alone vs. Placebo-Placebo
  * Ethanol Alone vs. Tasimelteon + Ethanol
  * Tasimelteon Alone vs. Placebo-Placebo
  * Tasimelteon Alone vs. Tasimelteon + Ethanol

SECONDARY OUTCOMES:
Pharmacokinetic parameters (AUC, Cmax, Tmax) of tasimelteon, tasimelteon's metabolites, and ethanol | Approximately Days 1, 8, 15, and 22: predose, 0.25, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours after dosing
Safety and tolerability as measured by spontaneous reporting of AEs, and clinically significant changes in laboratory parameters, ECG parameters, and vital signs | Screening (approximately Day -10), Days -2, -1, 1, and approximately Days 8, 15, 22, 23
The Columbia-Suicide Severity Rating Scale will be used to assess suicidal behavior and ideation. | once per day at Screening (approximately day -7),Day -1 (baseline), approximately Days 1, 8, 15, 22 and 23 (end of study)

CONTACTS AND LOCATIONS:
Locations (1):
- INC Research Toronto, Inc., Toronto, Ontario, Canada